CLINICAL TRIAL: NCT01159964
Title: Study of GSK2302032A Antigen-Specific Cancer Immunotherapeutic in Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: Evaluation of a New Anti-cancer Vaccine for Patients With Non-small Cell Lung Cancer, After Tumor Removal by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study termination due to negative Phase III of another study product from same technology platform.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113174
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Antigen-Specific Cancer Immunotherapeutic (ASCI); PRAME; PRAME-positive stage IB, II or IIIA Non-Small Cell Lung Cancer patients after complete surgical resection; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (3):
- Cohort 1 (Experimental): Subjects will receive investigational dose-level A (different from dose-levels B and C). All patients are to receive 13 injections of the immunotherapeutic GSK2302032A
  Interventions: Biological: Immunotherapeutic GSK2302032A, different formulations
- Cohort 2 (Experimental): Subjects will receive investigational dose-level B (different from dose-levels A and C). All patients are to receive 13 injections of the immunotherapeutic GSK2302032A
  Interventions: Biological: Immunotherapeutic GSK2302032A, different formulations
- Cohort 3 (Experimental): Subjects will receive investigational dose-level C (different from dose-levels A and B). All patients are to receive 13 injections of the immunotherapeutic GSK2302032A
  Interventions: Biological: Immunotherapeutic GSK2302032A, different formulations

INTERVENTIONS:
Biological: Immunotherapeutic GSK2302032A, different formulations — Intramuscular administration
  Other Names: PRAME ASCI

SUMMARY:
The purpose of this clinical study is to assess the safety and immunogenicity of the immunotherapeutic product GSK 2302032A when given to Non-Small Cell Lung Cancer (NSCLC) patients, after tumor removal by surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with completely resected (R0 resection), pathologically proven stage IB, II or IIIA NSCLC. Patients are allowed to receive adjuvant platinum-based chemotherapy for the treatment of the current NSCLC between surgery and enrolment.
2. Written informed consent for PRAME gene expression screening on resected tumor tissue has been obtained from the patient prior to shipment of the sample for expression testing, and written informed consent for the complete study participation has been obtained before the performance of any other protocol specific procedure.
3. Patient is >= 18 years of age at the time of signature of the first informed consent form.
4. The patient's tumor shows expression of the PRAME gene.
5. The surgical technique for resection of the patient's tumor is anatomical, involving at least a lobectomy or a sleeve lobectomy. The first ASCI administration will be given, either within 12 weeks after surgery or within 8 weeks after day 1 of last chemotherapy cycle and within 32 weeks after resection.
6. The patient is free of metastasis, as confirmed by a negative baseline computer tomogram (CT scan) of the chest and upper abdomen as well as CT scan or magnetic resonance imaging (MRI) of the brain. These tests are to be performed within 6 weeks for the CT scan of the chest and upper abdomen and within 12 weeks for the brain CT scan or MRI before first ASCI administration.
7. ECOG performance status of 0, 1 or 2.
8. Adequate bone-marrow reserve, renal, adrenal and hepatic function as assessed by standard laboratory criteria
9. Female patients of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal-ligation, hysterectomy, ovariectomy or post-menopause.
10. Female patient of childbearing potential may be enrolled in the study, if the patient:

    * has practiced adequate contraception for 30 days prior to study product administration, and
    * has a negative pregnancy test on the day of administration, and
    * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the study product administration series.
11. In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. The primary tumor was removed by segmentectomy or wedge resection.
2. The patient has received any anti-cancer specific treatment, including radiotherapy, immunotherapy, chemotherapy or neo-adjuvant chemotherapy, except for the treatment of previous malignancies allowed by the protocol.
3. The patient requires concomitant treatment (more than 7 consecutive days) with systemic corticosteroids or any other immunosuppressive agents.
4. Use of any investigational or non-registered product (drug or vaccine, except influenza vaccine in the context of H1N1 mass-vaccination) other than the study product within the 30 days preceding the first dose of study product, or planned use during the study period.
5. The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for more than 3 years and highly likely to have been cured.
6. History of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
7. History of confirmed adrenal dysfunction.
8. The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
9. The patient has received a major organ allograft.
10. The patient is known to be Human Immunodeficiency Virus (HIV) -positive.
11. The patient has an uncontrolled bleeding disorder.
12. The patient has uncontrolled congestive heart failure or uncontrolled hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia at the time of enrolment.
13. The patient needs home oxygenation.
14. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
15. The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
16. For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2011-10-19 (Actual); Study Completion 2014-09-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities during study treatment | During the study treatment period (up to 112 weeks, approximately 2 years and 2 months)
Occurrence of dose-limiting toxicities during study follow-up | 12 months after concluding visit (week 112)
Anti-PRAME humoral immune response | Assessed post-dose 4 (Week 12)
Anti-PRAME humoral immune response | Throughout the study (Day 0 until 12 months after concluding visit (week 112))

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) and serious adverse events | During the whole study treatment period until 30 days after the last treatment administration.
The anti-PRAME cellular (T-cell) response | At 6 defined time-points during the study (Week 0, 12, 24, 72 and 112) and follow-up period (6 months later).
The anti-PRAME humoral immunogenicity | At 10 defined timepoints during the study (Week 0, 6, 12, 24, 48, 72, 96, 112), and follow-up period (6 and 12 months later).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (7):
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Seattle, Washington
- France (4):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (10):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Italy (5):
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
- Poland (5):
  - GSK Investigational Site, Chęciny
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Zakopane
- Russia (4):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pujol JL, De Pas T, Rittmeyer A, Vallieres E, Kubisa B, Levchenko E, Wiesemann S, Masters GA, Shen R, Tjulandin SA, Hofmann HS, Vanhoutte N, Salaun B, Debois M, Jarnjak S, De Sousa Alves PM, Louahed J, Brichard VG, Lehmann FF. Safety and Immunogenicity of the PRAME Cancer Immunotherapeutic in Patients with Resected Non-Small Cell Lung Cancer: A Phase I Dose Escalation Study. J Thorac Oncol. 2016 Dec;11(12):2208-2217. doi: 10.1016/j.jtho.2016.08.120. Epub 2016 Aug 17. PMID 27544054
- See also: Results for study 113174 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113174?search=study&b%22b''%22#rs